CLINICAL TRIAL: NCT06534879
Title: The Effect of Psychosocial Factors on Academic Success in Physiotherapy and Rehabilitation Students
Brief Title: The Effect of Psychosocial Factors on Academic Success in University Students
Status: Not yet recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Muserrefe Nur Keles, Associate Professor, Gazi University
Other Study IDs: 88881925
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Students; Education
Keywords: University Student; Physicosocial factor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Psychological well-being is defined as the person fulfilling his/her potential in a completely good mood. It is seen as the result of a life lived well and is an important factor for students to adapt to university life. Psychological well-being includes dimensions such as self-acceptance, establishing positive relationships, autonomy, mastery of the environment, personal development and purpose in life. Students who have just started university have to adapt to a new learning model and the academic pressure on them is also increasing. This period of students' lives is considered to be one of the stages when anxiety is highest and psychological well-being is lowestThe examination of the potential predictive relationship between psychosocial factors and psychological goodness described earlier in a university student, provides a more holistic perspective for potential educators, researchers and health practitioners. Although the literature was examined, although the effects of some of the psychosocial factors on university students, physiotherapy and rehabilitation students have been found to have insufficient studies on the effect of psychosocial factors on academic success.

For this reason, in our study, physiotherapy and rehabilitation students will be evaluated with the level of empathy, self -esteem, social/emotional competence, mental good formation, situational/continuous anxiety (anxiety), motivation, satisfaction and loneliness surveys from life and the relationship between them and the academic achievements of the students will be investigated. .

DETAILED DESCRIPTION:
Psychological well-being is defined as the person fulfilling his/her potential in a completely good mood. It is seen as the result of a life lived well and is an important factor for students to adapt to university life. Psychological well-being includes dimensions such as self-acceptance, establishing positive relationships, autonomy, mastery of the environment, personal development and purpose in life. Students who have just started university have to adapt to a new learning model and the academic pressure on them is also increasing. This period of students' lives is considered to be one of the stages when anxiety is highest and psychological well-being is lowest. Some studies have already shown that the level of psychological well-being in university students is low. (2,3) Various models support possible psychosocial factors related to psychological well-being. From a general perspective, the psychoeducational approach is an integrative framework for the development and evaluation of psychological and educational constructs such as social skills, empathy, self-concept, anxiety and emotional intelligence, among others. More specific frameworks for the development of standards for high-quality professional education in psychology, such as the EuroPsy, include the following higher education competencies: adequate levels of empathy or anxiety, socially responsible attitudes, emotion management, problem solving and learning style preferences. Other frameworks, such as the European Higher Education Area and the Organisation for Economic Co-operation and Development, emphasise the importance of developing systemic competencies that include interpersonal and intrapersonal psychological resources such as emotional intelligence, self-esteem, social skills, social responsibility and empathy. From a psychological perspective, emotions are fundamental constructs related to psychological well-being and life satisfaction, according to classical theoretical models. Other more contemporary models include the models of Bisquerra and Pérez-Escoda. These models propose that emotional/psychological skills can be divided into two poles on a continuum. The positive side includes elements such as self-confidence, social skills and empathic attitudes, while the negative side includes symptoms such as anxiety. According to the existing empirical literature, both sides appear to be related to psychological well-being. The higher the satisfaction with the academic environment in general (content of university subjects, types of assessments used, methodologies applied to learning, teaching/learning styles, etc.), the greater the psychological well-being perceived by university students. Social skills are measured by the individual's general social competence and the interpersonal and intrapersonal strategies used. These skills appear to be related to academic performance in the university environment. Positive social relationships have been shown to be related to psychological well-being. On the positive side of the psychological continuum, emotional intelligence connects emotions with reason; in other words, just as our cognitive processes affect our emotional states, emotions affect our thoughts. The concept of emotional intelligence is defined as cognitive abilities that can be measured by tasks that involve the processing of emotional information. Recent research on emotional intelligence emphasizes the role of emotional intelligence in individuals' ability to adapt to their daily life environments and shows that emotional intelligence is linked to well-being. The effect of high emotional intelligence on academic performance in university students has been investigated and the role of emotional skills has been emphasized. Some authors have emphasized the importance of emotional intelligence as a type of psychosocial adaptation in the university education environment, as a possible predictor of psychological well-being. Several studies involving university students have examined the effect of adequate emotional intelligence skills on academic performance and have emphasized the key role of emotional skills. This shows the key role of emotional intelligence and its related dimensions (such as empathy) in university teaching and learning environments with students. Empathy is the ability that allows us to know how other people feel, what they think, understand their intentions, predict their behaviors and understand their emotions. Some studies on empathy have focused on analyzing empathy in young people because it contributes to the development of social skills and prosocial behaviors. It is seen that the psychological well-being perceived by students is strongly related to empathy. In a study conducted with a group of university students, Gustems Carnicer and Calderon found that students at high risk of psychological distress had higher scores in terms of empathic stress. They also found a direct relationship between psychological distress and emotional discharge, cognitive avoidance, alternative reward seeking and surrenderThey also found a direct relationship between psychological distress and emotional ejaculation, cognitive avoidance, search for alternative rewards and surrender. Recent research has reported the relationships between emotional ability known as empathy in university students and subjective well -being.

The concept of self is considered a complex term because of the difficulty of distinguishing from similar terms such as self -esteem. Many writers often call it the labels they give to them in relation to their bodies, behaviors and emotions. Behavioral, emotional and social functionality is explained by the perception of the individual's experiences; Therefore, the person's self -self -concept can be a procedure of the psychological good. In a study conducted with university students in the field of self -concept within the cooperation structure, it was seen that there was a development in the concept of self. Other studies have reported that there are positive relationships between psychological goodness and physical self -concept and self -esteem. For this reason, it is possible to include the concept of self as a possible factor associated with the psychological profiles of university students.

On the negative side of psychological continuity, anxiety is thought to be synonymous with other concepts such as stress, fear or distress. Spielberger et al. In addition to the activation of the autonomic nervous system, it defines anxiety as an emotional reaction that is externalized through tension, anxiety, irritability and anxiety. Spielberger, Gorsuch and Lushene reveal two types of anxiety depending on the length of time: situation and continuous anxiety. According to Spielberger, the state anxiety refers to an instant emotional state that can be changed over time, while continuous anxiety is a relatively stable tendency, tendency or personality trait. The concepts of different anxiety (situation and feature) need to be examined. The majority of the scientific literature suggest that approximately 50 %of university students experience significant anxiety. Research, which focuses on the university population, concluded that the effects of anxiety are closely related to some variables such as academic performance, quitting, psychological and emotional goodness. The examination of the potential predictive relationship between psychosocial factors and psychological goodness described earlier in a university student, provides a more holistic perspective for potential educators, researchers and health practitioners. Although the literature was examined, although the effects of some of the psychosocial factors on university students, physiotherapy and rehabilitation students have been found to have insufficient studies on the effect of psychosocial factors on academic success.

For this reason, in our study, physiotherapy and rehabilitation students will be evaluated with the level of empathy, self -esteem, social/emotional competence, mental good formation, situational/continuous anxiety (anxiety), motivation, satisfaction and loneliness surveys from life and the relationship between them and the academic achievements of the students will be investigated. .

ELIGIBILITY:
Inclusion Criteria:

* Being an active student in the physiotherapy and rehabilitation department
* willing to participate

Exclusion Criteria:

* not answering survey questions completely

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population of the study will consist of all students in the Department of Physiotherapy and Rehabilitation. The study aimed to reach the entire population without selecting a sample.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-08-05 (Estimated); Primary Completion 2024-08-25 (Estimated); Study Completion 2024-09-05 (Estimated)

PRIMARY OUTCOMES:
Rosenberg Self-Esteem Scale | 1 day
  The purpose of the 10 item RSE scale is to measure self-esteem. Originally the measure was designed to measure the self-esteem of high school students. However, since its development, the scale has been used with a variety of groups including adults, with norms available for many of those groups.
Empathy Assessment Scale | 1 day
  EAS is a valid and reliable measurement tool to assess the empathy levels of individuals in three dimensions: Social interaction, cognitive behavior, and emotional identification. EAS can be used to evaluate the empathy levels for research, education, and other interventional purposes.
State Trait Anxiety Inventory | 1 day
  The STAI is a validated 20 item self report assessment device which includes separate measures of state and trait anxiety. The original STAI form was constructed by Charles D. Spielberger, Richard L. Gorsuch, and Robert E. Lushene in 1964.
Satisfaction With Life Scale | 1 day
  The SWLS is a short 5-item instrument designed to measure global cognitive judgments of satisfaction with one's life. The scale usually requires only about one minute of a respondent's time, where respondents answer on a Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Muserrefe Nur Keles, PhD, Study Chair — Gazi University